CLINICAL TRIAL: NCT06242509
Title: Impact of Intestinal Enrichment in Akkermansia Muciniphila by Next-generation Hormonal Therapies on Castration Resistant-prostate Cancer Response
Brief Title: Intestinal Akkermansia Muciniphila in Prostate Cancer
Acronym: AkkPRO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221176
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic castration resistant prostate cancer (CRPC) receiving next generation hormonal therapy
  Interventions: Diagnostic Test: Biological samples

INTERVENTIONS:
Diagnostic Test: Biological samples — Plasma sampling ans stool sampling
  * at inclusion
  * at 1 month
  * at 3 months
  * at progression within the 3 months

SUMMARY:
Prostate cancer has the highest incidence and is the second leading cause of cancer death in men in western countries. Androgen deprivation therapy is the backbone treatment. However, after a latency hormone sensitive prostate cancer (HSPC) usually progresses to castration-resistant prostate cancer (CRPC) requiring treatments including next generation hormonal therapies with Abiraterone Acetate (AA). This, with limited survival.

A particularly challenging area of interest to improve outcome in cancer is the interaction between the microbiome and anti-cancer therapies. Emerging data demontrate in pre-clincal studies that prostate cancer alters the microbiota, with loss of diversity and depletion of beneficial bacteria including A. muciniphila. In the other hand, Androgen deprivation therapy, reverses these effects. Specifically, in advanced disease with castration-resistant prostate cancer (CRPC), it has been shown in small studies that Abiraterone Acetate, can modulate patient-associated gastro-intestinal microbiota through promoting the growth of A. muciniphila.

The goal of our study is to confirm that AA could promote fecal Akkermansia muciniphila growth and to use the enrichment of fecal Akkermansia muciniphila as a minimally invasive biomarker of response to AA in first line metastatic CRPC.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and not opposed to the study
* Be ≥ 18 years of age at the time of inclusion.
* Histologically or cytologically documented adenocarcinoma of the prostate.
* Have metastatic castration-resistant prostate cancer with castrate-level testosterone (<50 ng/dL) during the study
* Initiation of abiraterone acetate therapy or any other next-generation hormonal therapies within 15 days after inclusion
* Participants must be able and willing to comply with the study visit schedule and study procedures
* Affiliated with French social security

Exclusion Criteria:

* CRPC patients who were previously treated with any next generation hormonal therapies in a metastatic CRPC setting
* Person under legal protection
* Inability to obtain the non-opposition

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic CRPC receiving next generation hormonal therapy
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Relative abundance of Akkermansia muciniphila | At 1 month
  Between baseline and Month 1 of next-generation hormonotherapy (NGHT), compared between responders versus non-responders.
  The response is defined as an early PSA decrease > 50% at one month of NGHT.

SECONDARY OUTCOMES:
Relative variation of the relative abundance of Akkermansia muciniphila | At 3 months
  Between baseline and Month 3 of AA treatment, compared between responders versus non responders
Relative variation in PSA | At 1 month
  Relative variation in PSA between baseline PSA and nadir value, according to fecal Akkermansia muciniphila enrichment
Receiver Operating curve (ROC) | At 1 month
  Receiver Operating curve (ROC) of the baseline relative abundance of fecal Akkermansia muciniphila to predict PSA response
Receiver Operating curve (ROC) | At 3 months
  Receiver Operating curve (ROC) of the baseline relative abundance of fecal Akkermansia muciniphila to predict PSA response
PSA progression-free (PSA-PFS) survival | At 3 months
  According to fecal Akkermansia muciniphila baseline relative abundance. PSA-PFS will be defined as the time from treatment initiation to PSA progression as per PCWG3 (The Prostate Cancer Working Group 3) or death, whichever occurs first; patients without event at M3 will be treated as censored observations.
Anti- Akkermansia muciniphila IgG levels | At baseline
Anti- Akkermansia muciniphila IgG levels | At 1 month
Anti- Akkermansia muciniphila IgG levels | At 3 months
Anti- Akkermansia muciniphila IgA levels | At baseline
Anti- Akkermansia muciniphila IgA levels | At 1 month
Anti- Akkermansia muciniphila IgA levels | At 3 months
Alpha diversity | At baseline
  Assessed by Shannon index (Microbial Richness)
Alpha diversity | At 1 month
  Assessed by Shannon index (Microbial Richness)
Alpha diversity | At 3 months
  Assessed by Shannon index (Microbial Richness)
Beta diversity | At baseline
  Assessed by Bray-Curtis dissimilarity (Microbial Diversity)
Beta diversity | At 1 month
  Assessed by Bray-Curtis dissimilarity (Microbial Diversity)
Beta diversity | At 3 months
  Assessed by Bray-Curtis dissimilarity (Microbial Diversity)

IPD SHARING:
Plan to Share IPD: Undecided